CLINICAL TRIAL: NCT00864305
Title: A Relative Bioavailability Study of Gabapentin 400 mg Capsules Under Non-fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B-09237
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Gabapentin; Healthy subjects
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Gabapentin 400 mg capsules
  Interventions: Drug: Gabapentin 400 mg capsules; Drug: Gabapentin 400 mg capsules, single dose
- B (Active Comparator): Neurontin 400 mg capsules
  Interventions: Drug: NEURONTIN® 400 mg capsules

INTERVENTIONS:
Drug: Gabapentin 400 mg capsules — A: Experimental Subjects received Purepac formulated products under fed conditions
  Other Names: Gabapentin
  Arms: A
Drug: NEURONTIN® 400 mg capsules — B: Active comparator Subjects received Parke-Davis's marketed product
  Other Names: Gabapentin
  Arms: B
Drug: Gabapentin 400 mg capsules, single dose — C: Experimental Subjects received Purepac formulated products under fasting conditions
  Other Names: Gabapentin
  Arms: A

SUMMARY:
To compare the relative bioavailability of gabapentin 400 mg capsules (Purepac) with that of NEURONTIN® 400 mg capsules (Parke-Davis) in healthy adult male subjects under non-fasting conditions, and to compare the differences in plasma levels after dosing the test formulation with and without food

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Single dose, randomized, three-period, three-treatment, six-sequence crossover study under non-fasting conditions (test and reference) and fasting (test) conditions

Official Title: A relative Bioavailability Food Challenge Study of Gabapentin 400 mg Capsules

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* All subjects selected for this study will be males 18 to 45 (inclusive) years of age. Weight range of the subjects shall be 135-246 pounds, with individual weight variation not more than 10% ± from normal for height and body frame (Metropolitan Life, 1983, Height, Weight, Body Chart).
* Each subject shall be given a general physical examination within 21 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.

At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.

Adequate blood and urine samples should be obtained within 21 days before beginning of the first period and at the end of the trial for clinical laboratory measurements. Clinical laboratory measurements will include the following:

Hematology: hemoglobin, hematocrit, red blood cell count, platelets, and white blood cell count (with differential).

Clinical Chemistry: creatinine, BUN, glucose, SGOT, SGPT, bilirubin, and alkaline phosphate Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.

HTLV III Screen: (pre-study only) Hepatitis-B Surface Ag Screen: (pre-study only) Drugs of Abuse Screen: (pre-study only) Subjects will be selected if all above are normal.

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption, drug addition, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be restricted. If the clinical values are outside the range on testing, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* All subjects will have urine samples assayed for the presence of drugs of abuse as a part of the clinical laboratory screening procedures. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to starting the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the start of the study will not be allowed to participate.
* Subjects who have been exposed to known hepatic enzyme inducting or inhibiting agents within thirty (30) days prior to dosing will not be allowed to participate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1997-12; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Siler, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc, Saint Charles, Missouri, United States